CLINICAL TRIAL: NCT02733562
Title: The Effect of Different Eating Habits on Weight Loss in the First Year After Sleeve Gastrectomy
Brief Title: Results of Sleeve Gastrectomy Surgery in Relation With Eating Habits (After One Year)
Acronym: Behavior
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of the Department of Surgery, Assuta Medical Center
Other Study IDs: AMC 0216
Record Dates: First submitted 2016-03-26; First posted 2016-04-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Other Habit and Impulse Disorders; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Binge eaters: Classificated preoperatively
- Volume eaters: Classificated preoperatively
- sweet eaters: Classificated preoperatively
- snack eaters: Classificated preoperatively

SUMMARY:
Sleeve gastrectomy is one of the most common surgical procedures performed today for patients that undergo bariatric surgery. One of the primary reasons for morbid obesity is unhealthy eating habits and the belief that changes in those habits can ensure the success. Objectives: The investigators aimed to explore the effect of different eating habits prior to the bariatric surgery on the surgery success and on different aspect of quality of life. Design: The investigators conducted this study on patients that underwent sleeve gastrectomy as the first bariatric operation.

DETAILED DESCRIPTION:
The investigators conducted this study on patients that underwent sleeve gastrectomy as the first bariatric operation. The investigators divided the patients into groups according to their pre-operation eating habits: binge, sweet, snack and high volume and compared different aspects of the surgery such as weight loss, BMI and distance from ideal weight. The investigators also examined the effect of the surgery on the quality of life, sexual life, physical activity, eating habits and satisfaction from the surgery by a telephonic survey that was conducted up to one year after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity
* approved for bariatric surgery by the hospital's committee
* Patients that underwent primary surgery

Exclusion Criteria:

* recurrent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
weight loss | one year
  measured in KG

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nikiforova I, Barnea R, Azulai S, Susmallian S. Analysis of the Association between Eating Behaviors and Weight Loss after Laparoscopic Sleeve Gastrectomy. Obes Facts. 2019;12(6):618-631. doi: 10.1159/000502846. Epub 2019 Nov 20. PMID 31747668